CLINICAL TRIAL: NCT03511664
Title: VISION: An International, Prospective, Open Label, Multicenter, Randomized Phase 3 Study of 177Lu-PSMA-617 in the Treatment of Patients With Progressive PSMA-positive Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Study of 177Lu-PSMA-617 In Metastatic Castrate-Resistant Prostate Cancer
Acronym: VISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSMA-617-01; 2018-000459-41 (EudraCT Number); CAAA617A12301 (Other: Novartis)
Expanded Access: NCT04825652 (No longer available)
Record Dates: First submitted 2018-04-13; First posted 2018-04-30 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: Metastatic castration-resistant prostate cancer; mCRPC; 177Lu-PSMA-617; PSMA-617; PSMA-11; radioligand therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: Participants in the Main Study were randomized in a 2:1 ratio to receive either 177Lu-PSMA-617 plus BSC/BSoC or BSC/BSoC only. The sub-study was conducted in a non-randomized cohort (AAA617+ BSC/BSoC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC) (Experimental): Patients randomized to receive the investigational product received 7.4 GBq (+/- 10%) 177Lu-PSMA-617 intravenously every 6 weeks (+/- 1 week) for a maximum of 6 cycles. Best supportive/best standard of care (BS/BSOC) might be used
  Interventions: Drug: 177Lu-PSMA-617; Other: Best supportive/best standard of care
- Best supportive/best standard of care (BS/BSOC) alone (Other): Patients randomized to this arm received best supportive/best standard of care (BS/BSOC) as determined by the investigator
  Interventions: Other: Best supportive/best standard of care

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Administered intravenously once every 6 weeks (1 cycle) for a maximum of 6 cycles. After 4 cycles, patients were assessed for (1) evidence of response, (2) residual disease, and (3) tolerance to 177Lu-PSMA-617. If all 3 assessments were met the patient might received an additional 2 cycles of 177Lu-PSMA-617.
  Arms: 177Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC)
Other: Best supportive/best standard of care — Best supportive/best standard of care as defined by the local investigator

SUMMARY:
The primary objective of this study was to compare the two alternate primary endpoints of radiographic progression-free survival (rPFS) and overall survival (OS) in patients with progressive prostate-specific membrane antigen (PSMA)-positive metastatic castration-resistant prostate cancer (mCRPC) who received 177Lu-PSMA-617 in addition to best supportive/best standard of care (BSC/BSoC) versus patients treated with best supportive/best standard of care alone.

DETAILED DESCRIPTION:
The study for each participant consisted of a Screening period, a Treatment period and a Follow-up period.

Sub-study A dosimetry, PK and ECG sub-study was conducted in a non-randomized cohort (AAA617+BSC/BSoC) of 30 patients at sites in Germany to provide a more complete assessment of the safety aspects of AAA617. Aside from additional assessments to collect data for dosimetry, PK, urinary metabolites and ECG, patients in the sub-study were screened for eligibility, treated and followed up similarly to the AAA617+BSC/BSoC (investigational arm) patients in the main study.

Screening and randomization:

During the screening period of up to 28 days before starting randomized treatment, each participant was assessed for PSMA positivity by gallium (68Ga) gozetotide imaging PET/scan per the pre-defined read rules, by the Sponsor's central reader. Only patients with PSMA-positive metastatic PC and meeting all other inclusion/exclusion criteria were randomized in a 2:1 ratio to receive either 177Lu-PSMA-617 plus BSC/BSoC or BSC/BSoC only. Randomized patients were stratified on the following factors: LDH level (=< or > 260 UI/L), presence of liver metastases (Yes or No), eastern cooperative oncology group (ECOG) score (0-1 or 2) and inclusion of NAAD in the BSC/BSoC (at time of randomization (Yes or No)). Protocol- specified BSC/BSoC for each patient was initiated by the investigating physician prior to patient randomization and maintained throughout the study. On-study changes to BSC/BSoC were allowed and at the discretion of the investigating physician.

Randomized treatment:

"Randomized treatment" in this study refers to AAA617+BSC/BSoC (investigational arm) and BSC/BSoC only (control arm). For the sub-study, "study treatment" refers to AAA617+BSC/BSoC (also referred to as the investigational arm), as no randomization occurred in the sub-study. When discussing aspects of the study which are applicable to both the main and sub-study, the term 'randomized treatment' will be used throughout this document. The term 'study treatment' will be used only when specifically referring to the sub-study.

Patients randomized to the investigational arm began AAA617 dosing within 28 days of randomization. These patients received BSC/BSoC and 7.4 GBq (+/-10%) AAA617 once every 6 weeks (+/- 1 week) for a maximum of 6 cycles.

After the Cycle 4 treatment and prior to Cycle 5 treatment, the Investigator had to determine if:

* The patient showed evidence of response (i.e. radiological, PSA, clinical benefit)
* The patient had signs of residual disease on CT with contrast/MRI or bone scan
* The patient had shown good tolerance to the AAA617 treatment

If the patient met all of the criteria above and agreed to continue with additional treatment of AAA617 the investigator could administer a further 2 cycles. A maximum of 6 cycles of radioligand therapy was allowed. If the patient did not meet any of the criteria or did not agree to additional AAA617 treatment, then no additional doses of AAA617 were administered after Cycle 4. After the last cycle of AAA617, patients continued BSC/BSoC alone, as long as the investigator felt they were clinically benefiting or until they required a treatment regimen not allowed in this study. For both treatment arms, the cycle duration for Cycle 1-6 was 6 weeks and for Cycle 7 and beyond, 12 weeks. From Cycle 7 onwards, all patients from both treatment arms only received BSC/BSoC.

End of treatment:

An End of Treatment (EOT) visit was scheduled approximately 30 days after the last dose of AAA617 or the date of the BSC/BSoC end of treatment decision (whichever occurred later), but before the initiation of subsequent anti-cancer treatment, outside of what was allowed on study. Once a patient discontinued the randomized treatment part of the study for any reason, an EOT visit was scheduled.

Long-term follow-up:

Patients on the active part of the study at the time of the final analysis of OS had an EOT visit at the next planned visit after implementation of V5.0/5.1 of the protocol and moved into long-term follow-up, unless they specifically withdrew consent from long-term follow-up of the study.

Patients who consented to be followed for long-term status updates, entered the long-term follow-up period after the EOT visit. The long-term follow-up period included the collection of rPFS (if the patient discontinued for reasons other than radiographic progression), OS, information about new treatments along with the patient's response to these treatments, AE assessment, and results of hematology and chemistry testing. During the follow-up, patients were contacted every 3 months (+/-1 month) via phone, email, or letter until a long-term follow-up study became available, until death or until withdrawal of consent, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and sign an approved informed consent form (ICF).
2. Patients must have the ability to understand and comply with all protocol requirements.
3. Patients must be >= 18 years of age.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Patients must have a life expectancy >6 months.
6. Patients must have histological, pathological, and/or cytological confirmation of prostate cancer.
7. Patients must be 68Ga-PSMA-11 Positron Emission Tomography (PET)/Computed Tomography (CT) scan positive, and eligible as determined by the sponsor's central reader.
8. Patients must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
9. Patients must have received at least one NAAD (such as enzalutamide and/or abiraterone).
10. Patients must have been previously treated with at least 1, but no more than 2 previous taxane regimens. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a patient has received only 1 taxane regimen, the patient is eligible if: a. The patient's physician deems him unsuitable to receive a second taxane regimen (e.g. frailty assessed by geriatric or health status evaluation, intolerance, etc.).
11. Patients must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

    1. Serum/plasma PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 2.0 ng/mL.
    2. Soft-tissue progression defined as an increase >= 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions.
    3. Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan (2+2 PCWG3 criteria, Scher et al 2016).
12. Patients must have >= 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging obtained =< 28 days prior to beginning study therapy.
13. Patients must have recovered to =< Grade 2 from all clinically significant toxicities related to prior therapies (i.e. prior chemotherapy, radiation, immunotherapy, etc.).
14. Patients must have adequate organ function:

    a. Bone marrow reserve:
    * White blood cell (WBC) count >= 2.5 x 10^9/L (2.5 x 10^9/L is equivalent to 2.5 x 10^3/μL and 2.5 x K/μL and 2.5 x 10^3/cumm and 2500/μL) OR absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1.5 x 10^9/L is equivalent to 1.5 x 10^3/μL and 1.5 x K/μL and 1.5 x 10^3/cumm and 1500/μL)
    * Platelets >= 100 x 10^9/L (100 x 10^9/L is equivalent to 100 x 10^3/μL and 100 x K/μL and 100 x 10^3/cumm and 100,000/μL)
    * Hemoglobin >= 9 g/dL (9 g/dL is equivalent to 90 g/L and 5.59 mmol/L) b. Hepatic:
    * Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN). For patients with known Gilbert's Syndrome =< 3 x ULN is permitted
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3.0 x ULN OR =< 5.0 x ULN for patients with liver metastases c. Renal:
    * Serum/plasma creatinine =< 1.5 x ULN or creatinine clearance >= 50 mL/min
15. Albumin >3.0 g/dL (3.0 g/dL is equivalent to 30 g/L) [Inclusion #16 has been removed]

17. HIV-infected patients who are healthy and have a low risk of AIDS-related outcomes are included in this trial.

18. For patients who have partners of childbearing potential: Partner and/or patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principle investigator during the study and for 6 months after last study drug administration.

19. The best standard of care/ best supportive care options planned for this patient:

1. Are allowed by the protocol
2. Have been agreed to by the treating investigator and patient
3. Allow for the management of the patient without 177Lu-PSMA-617

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed.
2. Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 28 days prior to day of randomization.
3. Any investigational agents within 28 days prior to day of randomization.
4. Known hypersensitivity to the components of the study therapy or its analogs.
5. Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
6. Transfusion for the sole purpose of making a subject eligible for study inclusion.
7. Patients with a history of Central Nervous System (CNS) metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast).
8. A superscan as seen in the baseline bone scan.
9. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
10. Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
11. Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, patients with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible, as are patients with adequately treated non-melanoma skin cancer, superficial bladder cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 861 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (88):
- United States (45):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California Los Angeles, Nuclear Medicine, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Washington DC VA Medical Center, Nuclear Medicine Service, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Iowa City VA Medical Center, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane Medical Center, Tulane Cancer Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Chesapeake Urology Associates (CUA) P.A., Towson, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - VA St. Louis Health Care System - John Cochran, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Twain Office, Las Vegas, Nevada
  - Regional Cancer Care Associates, Central Jersey Division, East Brunswick, New Jersey
  - New Mexico Oncology Hematology Consultants Ltd., New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Duke Cancer Center, Durham, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Oregon Health and Science University, Nuclear Medicine, Portland, Oregon
  - Pennsylvania Cancer Specialists & Research Institute, Gettysburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - VA North Texas Health Care System, Nuclear Medicine Service, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Excel Diagnostics & Nuclear Oncology Center, Houston, Texas
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute Research, Seattle, Washington
- Belgium (3):
  - Jules Bordet Institute, Brussels
  - Saint Luc University Hospital, Brussels
  - University Hospitals Leuven, Campus Gasthuisberg, Department of Nuclear Medicine, Leuven
- Canada (7):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - London Health Sciences Centre, Division of Nuclear Medicine, London, Ontario
  - Ottawa Hospital, Cancer Center, Ottawa, Ontario
  - Sunnybrook Research Institute, Odette Cancer Center, Toronto, Ontario
  - CHUM - University Hospital of Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU of Quebec - Laval University, Québec
- Denmark (3):
  - Aalborg University Hospital, Oncology Department, Aalborg
  - Aarhus University Hospital, Department of Oncology, Aarhus
  - Rigshospitalet - University Hospital Copenhagen, Department of Oncology, Copenhagen
- France (7):
  - Bergonie Institute, Bordeaux
  - Center Jean Perrin, Clermont-Ferrand
  - Leon Berard Center, Lyon
  - Saint-Louis Hospital, Paris
  - Tenon Hospital, Paris
  - Institute Claudius Regaud, Toulouse Cancer Research Center, Toulouse
  - Gustave Roussy Oncology Institute, Villejuif
- Germany (4):
  - University Hospital Essen, Clinic for Nuclear Medicine, Essen
  - Hospital rechts der Isar, Department of Nuclear Medicine, Munich
  - University Hospital Muenster, Department of Nuclear Medicine, Münster
  - Rostock University Medical Center, Clinic and Polyclinic for Nuclear Medicine, Rostock
- Netherlands (4):
  - The Netherlands Cancer Institute, Amsterdam
  - St. Antonius Hospital, Nieuwegein
  - Radboud University Medical Center (Radboudumc), Nijmegen
  - UMC Utrecht, Utrecht
- VA Caribbean Healthcare System, San Juan, Puerto Rico
- Sweden (5):
  - Sahlgrenska University Hospital, Department of Oncology, Gothenburg
  - Skane University Hospital - Barngatan, Clinical Trials Unit, Lund
  - Karolinska University Hospital, Stockholm
  - Norrlands University Hospital, Cancer Center, Umeå
  - Uppsala University Hospital, Department of Oncology, Uppsala
- United Kingdom (9):
  - Bristol Hematology & Oncology Center, Bristol
  - Beatson West of Scotland Cancer Center, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Guy's Hospital, London
  - Royal Free Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Iravani A, Violet J, Azad A, Hofman MS. Lutetium-177 prostate-specific membrane antigen (PSMA) theranostics: practical nuances and intricacies. Prostate Cancer Prostatic Dis. 2020 Mar;23(1):38-52. doi: 10.1038/s41391-019-0174-x. Epub 2019 Oct 8. PMID 31595044
- [Result] Chi KN, Yip SM, Bauman G, Probst S, Emmenegger U, Kollmannsberger CK, Martineau P, Niazi T, Pouliot F, Rendon R, Hotte SJ, Laidley DT, Saad F. 177Lu-PSMA-617 in Metastatic Castration-Resistant Prostate Cancer: A Review of the Evidence and Implications for Canadian Clinical Practice. Curr Oncol. 2024 Mar 7;31(3):1400-1415. doi: 10.3390/curroncol31030106. PMID 38534939
- [Result] Fizazi K, Herrmann K, Krause BJ, Rahbar K, Chi KN, Morris MJ, Sartor O, Tagawa ST, Kendi AT, Vogelzang N, Calais J, Nagarajah J, Wei XX, Koshkin VS, Beauregard JM, Chang B, Ghouse R, DeSilvio M, Messmann RA, de Bono J. Health-related quality of life and pain outcomes with [177Lu]Lu-PSMA-617 plus standard of care versus standard of care in patients with metastatic castration-resistant prostate cancer (VISION): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 Jun;24(6):597-610. doi: 10.1016/S1470-2045(23)00158-4. PMID 37269841
- [Result] Herrmann K, Rahbar K, Eiber M, Sparks R, Baca N, Krause BJ, Lassmann M, Jentzen W, Tang J, Chicco D, Klein P, Blumenstein L, Basque JR, Kurth J. Renal and Multiorgan Safety of 177Lu-PSMA-617 in Patients with Metastatic Castration-Resistant Prostate Cancer in the VISION Dosimetry Substudy. J Nucl Med. 2024 Jan 2;65(1):71-78. doi: 10.2967/jnumed.123.265448. PMID 38050121
- [Result] Kuo PH, Yoo DC, Avery R, Seltzer M, Calais J, Nagarajah J, Weber WA, Fendler WP, Hofman MS, Krause BJ, Brackman M, Kpamegan E, Ghebremariam S, Benson T, Catafau AM, Kendi AT. A VISION Substudy of Reader Agreement on 68Ga-PSMA-11 PET/CT Scan Interpretation to Determine Patient Eligibility for 177Lu-PSMA-617 Radioligand Therapy. J Nucl Med. 2023 Aug;64(8):1259-1265. doi: 10.2967/jnumed.122.265077. Epub 2023 May 25. PMID 37230533
- [Result] Sartor O, de Bono J, Chi KN, Fizazi K, Herrmann K, Rahbar K, Tagawa ST, Nordquist LT, Vaishampayan N, El-Haddad G, Park CH, Beer TM, Armour A, Perez-Contreras WJ, DeSilvio M, Kpamegan E, Gericke G, Messmann RA, Morris MJ, Krause BJ; VISION Investigators. Lutetium-177-PSMA-617 for Metastatic Castration-Resistant Prostate Cancer. N Engl J Med. 2021 Sep 16;385(12):1091-1103. doi: 10.1056/NEJMoa2107322. Epub 2021 Jun 23. PMID 34161051
- [Result] Armstrong AJ, Sartor O, de Bono J, Chi K, Fizazi K, Krause BJ, Herrmann K, Rahbar K, Tagawa ST, Saad F, Beer TM, Wu J, Mirante O, Morris MJ. Association of Declining Prostate-specific Antigen Levels with Clinical Outcomes in Patients with Metastatic Castration-resistant Prostate Cancer Receiving [177Lu]Lu-PSMA-617 in the Phase 3 VISION Trial. Eur Urol. 2024 Dec;86(6):552-562. doi: 10.1016/j.eururo.2024.08.021. Epub 2024 Sep 5. PMID 39242323
- [Result] Chi KN, Armstrong AJ, Krause BJ, Herrmann K, Rahbar K, de Bono JS, Adra N, Garje R, Michalski JM, Kempel MM, Fizazi K, Morris MJ, Sartor O, Brackman M, DeSilvio M, Wilke C, Holder G, Tagawa ST. Safety Analyses of the Phase 3 VISION Trial of [177Lu]Lu-PSMA-617 in Patients with Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2024 Apr;85(4):382-391. doi: 10.1016/j.eururo.2023.12.004. Epub 2024 Jan 6. PMID 38185538
- [Result] Herrmann K, Gafita A, de Bono JS, Sartor O, Chi KN, Krause BJ, Rahbar K, Tagawa ST, Czernin J, El-Haddad G, Wong CC, Zhang Z, Wilke C, Mirante O, Morris MJ, Fizazi K. Multivariable models of outcomes with [177Lu]Lu-PSMA-617: analysis of the phase 3 VISION trial. EClinicalMedicine. 2024 Oct 4;77:102862. doi: 10.1016/j.eclinm.2024.102862. eCollection 2024 Nov. PMID 39430616
- [Result] Kuo PH, Morris MJ, Hesterman J, Kendi AT, Rahbar K, Wei XX, Fang B, Adra N, Garje R, Michalski JM, Chi K, de Bono J, Fizazi K, Krause B, Sartor O, Tagawa ST, Ghebremariam S, Brackman M, Wong CC, Catafau AM, Benson T, Armstrong AJ, Herrmann K. Quantitative 68Ga-PSMA-11 PET and Clinical Outcomes in Metastatic Castration-resistant Prostate Cancer Following 177Lu-PSMA-617 (VISION Trial). Radiology. 2024 Aug;312(2):e233460. doi: 10.1148/radiol.233460. PMID 39162634
- [Result] Morris MJ, de Bono J, Nagarajah J, Sartor O, Wei XX, Nordquist LT, Koshkin VS, Chi KN, Krause BJ, Herrmann K, Rahbar K, Vickers A, Mirante O, Ghouse R, Fizazi K, Tagawa ST. Correlation analyses of radiographic progression-free survival with clinical and health-related quality of life outcomes in metastatic castration-resistant prostate cancer: Analysis of the phase 3 VISION trial. Cancer. 2024 Oct 15;130(20):3426-3435. doi: 10.1002/cncr.35438. Epub 2024 Jun 21. PMID 39031642
- [Derived] Sundlov A, Sjogreen-Gleisner K. Peptide Receptor Radionuclide Therapy - Prospects for Personalised Treatment. Clin Oncol (R Coll Radiol). 2021 Feb;33(2):92-97. doi: 10.1016/j.clon.2020.10.020. Epub 2020 Nov 12. PMID 33189510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 86 sites across 9 countries. Belgium (3); Canada (7); Denmark (3); France (6); Netherlands (4); Sweden (5); UK (9); US (45); Germany (4, for the sub-study only).
Groups:
- Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC): Patients randomized to receive the investigational product received 7.4 GBq (+/- 10%) 177Lu-PSMA-617 intravenously every 6 weeks (+/- 1 week) for a maximum of 6 cycles. Best supportive/best standard of care (BS/BSOC) might be used
- Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone: Patients randomized to this arm received best supportive/best standard of care (BS/BSOC) as determined by the investigator
- Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC): non-randomized cohort (AAA617+ BS/BSOC) at sites in Germany to provide a more complete assessment of the safety aspects of AAA617. Patients were treated and followed up similarly to the AAA617+BSC/BSOC (investigational arm) patients in the main study
Period: Overall Study
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC)
Started (All randomized patients were included in the Full Analysis Set (FAS). Patients were included in the treatment arm to which they were randomized regardless of actual treatment received.) | 551 | 280 | 30
FAS Safety Analysis Set (The subset of patients in the Full Analysis Set (FAS) who received at least one dose of randomized treatment.) | 529 | 205 | 30
Progression-Free Survival (PFS) Full Analysis Set (PFS-FAS) (All patients randomized on or after 05-Mar-2019. Patients were included in the treatment arm to which they were randomized regardless of actual treatment received.) | 385 | 196 | 0
Response Evaluable Analysis Set (The subset of patients in the PFS-FAS with evaluable disease by RECIST at baseline. Patients were included in the treatment arm to which they were randomized.) | 319 | 120 | 0
Completed | 28 | 6 | 4
Not Completed | 523 | 274 | 26
Not completed — Death | 457 | 201 | 21
Not completed — Withdrew consent | 40 | 63 | 3
Not completed — Other protocol pre-specified reasons for discontinuation | 15 | 4 | 2
Not completed — Lost to Follow-up | 8 | 5 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Patient non-compliance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Total
Number analyzed (Participants) | 551 | 280 | 30 | 861
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 145 | 60 | 12 | 217
  ≥ 65-84 years | 398 | 214 | 18 | 630
  ≥ 85 years | 8 | 6 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 551 | 280 | 30 | 861
Race/Ethnicity, Customized [Number; unit: Participants] — Race 'Other' included Native Hawaiian or Other Pacific Islander, American Indian or Alaska Native and more than one race reported.
  Participants
    White | 486 | 235 | 30 | 751
    Black or African American | 34 | 21 | 0 | 55
    Asian | 9 | 11 | 0 | 20
    Other | 2 | 0 | 0 | 2
    Missing | 20 | 13 | 0 | 33

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Radiographic progression-free survival (rPFS) was defined as the time (in months) from the date of randomization to the date of radiographic disease progression based on the central review assessment per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria or death due to any cause. Patients who were alive without radiographic progression at the analysis data cut-off were censored for rPFS at the time of their last evaluable radiographic assessment. Date of censoring for rPFS: 1) The censoring date was the date when the last evaluable radiographic assessment (CT/MRI/bone scan) determined a lack of progression; 2) If there were no evaluable assessments, censoring occurred at the date of randomization; 3) Patients who had 2 or more consecutive missed tumor assessments immediately prior to PD or death were censored at the date of the last evaluable tumor assessment prior to those missing tumor assessments.
Time Frame: From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Median (99.2% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Months | 8.7 [7.9 to 10.8] | 3.4 [2.4 to 4.0]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Log Rank; one-sided stratified log-rank test; Hazard Ratio (HR) = 0.40, 99.2% CI 2-sided [0.29 to 0.57]

2. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time (in months) from the date of randomization to the date of death due to any cause. If the patient was not known to have died, then OS was censored. The censoring date was date of the last study visit, or contact, until the cut-off date. The cut-off date was not used for last contact date, unless the patient was seen or contacted on that date.
  Final OS was analyzed at the time of Primary analysis (Primary Analysis cut-off date = 27-Jan-2021) and an updated descriptive analysis of OS was re-run at the time of final analysis (Final Analysis cut-off date 14-Dec-2023).
Time Frame: From date of randomization until date of death from any cause, assessed up to 32 months (Primary Analysis cut-off date = 27-Jan-2021) and up to 66 months (Final Analysis cut-off date = 14-Dec-2023)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 551 | 280
Months
  Primary OS Analysis | 15.3 [14.2 to 16.9] | 11.3 [9.8 to 13.5]
  Final OS analysis | 15.3 [14.2 to 16.9] | 11.5 [9.9 to 13.5]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Primary OS Analysis; Test type: Superiority; p < 0.001, Log Rank; one-sided stratified log-rank test; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.52 to 0.74]
Statistical Analysis 2: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Final OS analysis; Test type: Superiority; Cox Proportional Hazard = 0.68, 95% CI 2-sided [0.58 to 0.81] — Cox PH model stratified by LDH (≤260 vs. >260 IU/L), liver metastases (yes/no), ECOG score (0-1 vs. 2), and NAAD inclusion in best supportive care at randomization (yes/no). IRT data used for stratification

3. Secondary Outcome: Number of Participants With Randomized/Study Treatment-emergent Adverse Events (TEAE)
Description: In the Main Study, "randomized treatment" refers to the investigational arm (AAA617+BSC/BSoC) and the control arm (BSC/BSoC). In the sub-study, "study treatment" refers to the investigational arm (AAA617+BSC/BSoC) without randomization:
  1. A randomized treatment-emergent adverse event (TEAE) is any adverse event that occurs from the start of randomized treatment to 30 days after the last administration of randomized treatment or prior to the initiation of subsequent anticancer treatment.
  2. A study treatment-emergent adverse event (TEAE) is any adverse event that occurs from the start of study treatment to 30 days after the last administration of study treatment or prior to the initiation of subsequent anticancer treatment.
  The distribution of randomized/study treatment-emergent adverse events (TEAEs) was done via the analysis of frequencies for TEAEs and Serious Adverse Event (TESAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From randomization till 30 days safety follow-up, assessed up to 66 months (Final Analysis cut-off date = 14-Dec-2023)
Population: FAS Safety Analysis Set. A patient with multiple grades for an AE is only counted under the maximum grade. Drug-related is related to any study drug (177Lu-PSMA-617 or BSC/BSoC). Study treatment refers to 177Lu-PSMA-617+BSC/BSoC.
Measure: Number; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC)
Number analyzed (Participants) | 529 | 205 | 30
Participants
  TEAE | 518 | 170 | 30
  Serious TEAE | 195 | 58 | 9
  Grade 3/4/5 TEAE | 284 | 79 | 11
  Drug-related TEAE | 451 | 59 | 19
  Serious Drug-related TEAE | 51 | 5 | 2
  Drug-related grade 3/4/5 TEAE | 152 | 8 | 6
  TEAE leading to reduction of 177Lu-PSMA-617 | 30 | 0 | 2
  TEAE leading to reduction of BSC/BSoC | 17 | 7 | 1
  TEAE leading to interruption of 177Lu-PSMA-617 | 85 | 2 | 4
  TEAE leading to interruption of BSC/BSoC | 50 | 14 | 1
  TEAE leading to discontinuation of 177Lu-PSMA-617 | 63 | 1 | 2
  TEAE leading to discontinuation of BSC/BSoC | 47 | 16 | 0
  Fatal TEAE | 19 | 6 | 2

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with evaluable disease at baseline per central review assessment.
Time Frame: as for outcome 1
Population: Response Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 319 | 120
Participants | 95 | 2
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Chi-squared; Two-sided Wald's Chi-square test (stratified); Odds Ratio (OR) = 24.99, 95% CI 2-sided [6.05 to 103.24]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1 per central review assessment.
Time Frame: as for outcome 1
Population: Response Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 319 | 120
Participants | 284 | 80
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Chi-squared; Two-sided Wald's Chi-square test (stratified); Odds Ratio (OR) = 5.79, 95% CI 2-sided [3.18 to 10.55]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause as per central review assessment.
Time Frame: From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS Full Analysis Set (PFS-FAS). Only participants for whom BOR was CR or PR and evaluable Duration of Response events (Progression or Death) included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 95 | 2
Months | 9.8 [9.1 to 11.7] | 10.6 [NA to NA] — NA: not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: Time to first Symptomatic Skeletal Event (SSE) was defined as the time (in months) from the date of randomization to the date of the SSE or death from any cause. The SSE date was the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever occurred first. SSE data for this endpoint were collected up through EOT visit. The censoring date was date of the last study visit (on or before the EOT visit).
Time Frame: as for outcome 1
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Months | 11.5 [10.3 to 13.2] | 6.8 [5.2 to 8.5]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Log Rank; Two-sided stratified log-rank test; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.40 to 0.62]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time (in months) from the date of randomization to the date of first evidence of radiographic, clinical or PSA progression or death due to any cause, whichever occurred first.
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Months | 5.9 [5.2 to 6.6] | 2.4 [2.2 to 3.0]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Log Rank; Two-sided stratified log-rank test; Cox Proportional Hazard = 0.30, 95% CI 2-sided [0.24 to 0.38]

9. Secondary Outcome: Best Percentage Change From Baseline in Prostate-specific Antigen (PSA) Level
Description: Best percentage change from baseline in PSA level was defined as the maximum percent decrease at any time post-baseline, including only patients with a baseline value and at least one non-missing post-baseline value (scheduled and unscheduled).
Time Frame: From date of randomization till 30 days safety fup, assessed up to approximately 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS Full Analysis Set (PFS-FAS). Only participants with evaluable post-baseline and baseline samples were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 333 | 138
Percentage change | -20.9 (142.6) | 50.4 (118.4)

10. Secondary Outcome: Percentage of Participants Achieving Prostate-specific Antigen (PSA) Response
Description: PSA response was defined as the proportion of patients who had a >= 50% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Percentage of participants | 46.0 [40.9 to 51.1] | 7.1 [4.0 to 11.7]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Chi-squared; Two-sided Wald's Chi-square test (stratified); Odds Ratio (OR) = 11.19, 95% CI 2-sided [6.3 to 20.0]

11. Secondary Outcome: Prostate-specific Antigen 80 (PSA80) Response
Description: PSA80 response was defined as the proportion of participants who had a >= 80% decrease in PSA from baseline confirmed by a PSA measurement >= 4 weeks later.
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Percentage of participants | 33.0 [28.3 to 37.9] | 2.0 [0.6 to 5.1]
Statistical Analysis 1: Comparison: Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) vs Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone; Test type: Superiority; p < 0.001, Chi-squared; Two-sided Wald's Chi-square test (stratified); Odds Ratio (OR) = 23.6, 95% CI 2-sided [8.6 to 65.1]

12. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response was defined as the duration between the date of first document PSA response (i.e. >= 50% decrease in PSA from Baseline) and the earliest date of PSA progression, where date of PSA progression was defined as: 1) Where a decline from baseline was documented, date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained at least 3 weeks later. Rises in PSA within the first 12 weeks of the date of first dose of randomized treatment were ignored; 2) Where no decline from baseline was documented, PSA progression was defined as a >= 25% increase from the baseline value along with an increase in absolute value of 2 ng/mL or more after 12 weeks from the date of first dose of randomized treatment (without confirmation) as specified in the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines.
Time Frame: From date of first documented PSA response till 30 days safety fup, assessed up to approximately 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS Full Analysis Set (PFS-FAS). Only participants with PSA progression were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 177 | 14
Months | 8.9 [7.6 to 10.7] | 4.4 [2.6 to 10.8]

13. Secondary Outcome: Best Percentage Change From Baseline in Alkaline Phosphatase (ALP) Level
Description: Best percentage change from baseline in alkaline phosphatase (ALP) level was defined as the maximum percent decrease at any time post-baseline, including only patients with a baseline value and at least one non-missing post-baseline value (scheduled and unscheduled).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 372 | 172
Percentage change | -14.4 (46.3) | 0.6 (33.8)

14. Secondary Outcome: Best Percentage Change From Baseline in Lactate Dehydrogenase (LDH) Level
Description: Best percentage change from baseline in lactate dehydrogenase (LDH) level was defined as the maximum percent decrease at any time post-baseline, including only patients with a baseline value and at least one non-missing post-baseline value (scheduled and unscheduled).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 371 | 168
Percentage change | -23.1 (23.8) | -9.2 (28.2)

15. Secondary Outcome: Time to Worsening in BPI-SF Pain Intensity Scale
Description: Time to worsening in BPI-SF pain intensity scale was defined as the time from randomization to the first occurring of an increase of worsening threshold (>=30% of baseline or >=2-point increase) at any time up through EOT visit compared to baseline, clinical disease progression, or death.
Time Frame: From date of randomization until date of End of Treatment (EoT), assessed up to 32 months (Primary Analysis cut-off date = 27-Jan-2021)
Population: PFS-Full analysis set. Only participants with evaluable events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 328 | 166
Months | 5.9 [4.8 to 6.9] | 2.2 [1.8 to 2.8]

16. Secondary Outcome: Time to Improvement After Worsening in BPI-SF Pain Intensity Scale
Description: Time to improvement after worsening in BPI-SF pain intensity scale was defined as the time from worsening of Pain Intensity score to a Pain Intensity score <= baseline.
Time Frame: as for outcome 15
Population: PFS-Full analysis set. Only participants with evaluable events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 144 | 76
Months | 2.8 [1.9 to 4.2] | 4.2 [2.8 to 11.3]

17. Secondary Outcome: Time to Worsening in BPI-SF Pain Interference Scale
Description: Time to worsening in BPI-SF pain interference scale was defined as the time from randomization to the first occurring of 1) an increase of worsening threshold (>=30% of baseline or >=2-point increase) at any time up through EOT visit compared to baseline, 2) clinical disease progression, or 3) death.
Time Frame: as for outcome 15
Population: PFS-Full analysis set. Only participants with evaluable events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 330 | 166
Months | 5.0 [4.2 to 6.1] | 2.3 [1.7 to 2.9]

18. Secondary Outcome: Time to Improvement After Worsening in BPI-SF Pain Interference Scale
Description: Time to improvement after worsening in BPI-SF pain interference scale was defined as the time from worsening of Pain Interference score to a Pain Interference score <= baseline.
Time Frame: as for outcome 15
Population: PFS-Full analysis set. Only participants with evaluable events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 176 | 72
Months | 3.0 [2.8 to 4.4] | 2.8 [1.7 to NA] — NA: not estimable due the number of censored participants at the time the analysis cut-off date was reached.

19. Secondary Outcome: Time to Worsening in BPI-SF Worst Pain Intensity Scale (Time to Disease Related Pain)
Description: Time to worsening in BPI-SF worst pain intensity scale (time to disease related pain) was defined as the time from randomization to the first occurring of worsening exceeding the threshold threshold (>=30% of baseline or >=2 point increase) at any time up through EOT visit compared to baseline, clinical disease progression, or death.
Time Frame: as for outcome 15
Population: PFS-Full analysis set. Only participants with evaluable events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 332 | 169
Months | 5.0 [4.2 to 5.9] | 2.0 [1.7 to 2.2]

20. Secondary Outcome: Change From Baseline in BPI-SF (Brief-Pain Inventory - Short Form) Pain Intensity Scale
Description: The BPI-SF is a generic pain assessment tool used in research and practice for pain assessment in musculoskeletal conditions. The higher the BPI-SF score, the worse the pain. The BPI-SF consists of 4 questions regarding pain intensity (worst pain intensity, least pain intensity, average pain intensity and pain right now), 2 questions on the use of analgesics, and 7 questions on how the level pain has interfered with the subject's life (General Activity, Mood, Walking Ability, Normal Work, Relations with other people, Sleep, Enjoyment of Life). Intensity items consist of an 11-response rating scale scored from 0 ("No Pain") to 10 ("Pain As Bad As You Can Imagine"). BPI-SF Pain intensity is the mean of non-missing items of the 4 individual scales, if there are 3 or more items not missing; otherwise this scale is set to missing.
Time Frame: Baseline (BL), Cycle 2 to Cycle 13 (Week 1 Day 1), End of Treatment (EoT) (cycle duration for Cycle 1-6 = 6 weeks and for Cycle 7 and beyond = 12 weeks)
Population: PFS Full Analysis Set (PFS-FAS). Only participants with non-missing score both at Baseline and at post-baseline visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Score on a scale
  Cycle 2, Week 1, Day 1 change from BL: number analyzed (Participants) | 311 | 100
  Cycle 2, Week 1, Day 1 change from BL | -0.59 (2.037) | 0.21 (2.404)
  Cycle 3, Week 1, Day 1 change from BL: number analyzed (Participants) | 274 | 52
  Cycle 3, Week 1, Day 1 change from BL | -0.62 (1.924) | 0.02 (2.033)
  Cycle 4, Week 1, Day 1 change from BL: number analyzed (Participants) | 223 | 32
  Cycle 4, Week 1, Day 1 change from BL | -0.42 (2.017) | 0.26 (2.383)
  Cycle 5, Week 1, Day 1 change from BL: number analyzed (Participants) | 183 | 21
  Cycle 5, Week 1, Day 1 change from BL | -0.49 (1.957) | 0.55 (3.144)
  Cycle 6, Week 1, Day 1 change from BL: number analyzed (Participants) | 162 | 13
  Cycle 6, Week 1, Day 1 change from BL | -0.41 (1.897) | 0.10 (2.740)
  Cycle 7, Week 1, Day 1 change from BL: number analyzed (Participants) | 123 | 11
  Cycle 7, Week 1, Day 1 change from BL | -0.48 (2.011) | -0.32 (1.585)
  Cycle 8, Week 1, Day 1 change from BL: number analyzed (Participants) | 86 | 5
  Cycle 8, Week 1, Day 1 change from BL | -0.18 (1.759) | -1.10 (2.205)
  Cycle 9, Week 1, Day 1 change from BL: number analyzed (Participants) | 55 | 6
  Cycle 9, Week 1, Day 1 change from BL | -0.70 (2.157) | 0.13 (1.780)
  Cycle 10, Week 1, Day 1 change from BL: number analyzed (Participants) | 33 | 2
  Cycle 10, Week 1, Day 1 change from BL | 0.02 (1.513) | 0.50 (1.768)
  Cycle 11, Week 1, Day 1 change from BL: number analyzed (Participants) | 12 | 2
  Cycle 11, Week 1, Day 1 change from BL | -0.40 (0.956) | 0.75 (1.768)
  Cycle 12, Week 1, Day 1 change from BL: number analyzed (Participants) | 4 | 0
  Cycle 12, Week 1, Day 1 change from BL | -1.00 (0.354) |
  Cycle 13, Week 1, Day 1 change from BL: number analyzed (Participants) | 1 | 0
  Cycle 13, Week 1, Day 1 change from BL | -0.75 (NA) — NA: Only one participant analyzed |
  End of Treatment (EoT) change from BL: number analyzed (Participants) | 165 | 88
  End of Treatment (EoT) change from BL | 0.46 (2.415) | 0.50 (2.405)

21. Secondary Outcome: Change From Baseline in BPI-SF (Brief-Pain Inventory - Short Form) Pain Interference Scale
Description: The BPI-SF is a generic pain assessment tool used in research and practice for pain assessment in musculoskeletal conditions. The higher the BPI-SF score, the worse the pain. The BPI-SF consists of 4 questions regarding pain intensity (worst pain intensity, least pain intensity, average pain intensity and pain right now), 2 questions on the use of analgesics, and 7 questions on how the level pain has interfered with the subject's life (General Activity, Mood, Walking Ability, Normal Work, Relations with other people, Sleep, Enjoyment of Life). Interference items consist of scores from 0 ("Does Not Interfere") to 10 ("Completely Interferes"). BPI-SF Interference scale is the mean of non-missing items of the 7 items on pain interference, if there are 4 or more items not missing; otherwise this scale is set to missing.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Score on a scale
  Cycle 2, Week 1, Day 1 change from BL: number analyzed (Participants) | 311 | 100
  Cycle 2, Week 1, Day 1 change from BL | -0.40 (2.167) | 0.58 (2.700)
  Cycle 3, Week 1, Day 1 change from BL: number analyzed (Participants) | 274 | 52
  Cycle 3, Week 1, Day 1 change from BL | -0.35 (2.348) | -0.15 (2.216)
  Cycle 4, Week 1, Day 1 change from BL: number analyzed (Participants) | 223 | 32
  Cycle 4, Week 1, Day 1 change from BL | -0.33 (2.249) | 0.21 (2.762)
  Cycle 5, Week 1, Day 1 change from BL: number analyzed (Participants) | 183 | 21
  Cycle 5, Week 1, Day 1 change from BL | -0.32 (2.223) | 0.52 (3.480)
  Cycle 6, Week 1, Day 1 change from BL: number analyzed (Participants) | 161 | 13
  Cycle 6, Week 1, Day 1 change from BL | -0.28 (2.166) | 0.49 (3.354)
  Cycle 7, Week 1, Day 1 change from BL: number analyzed (Participants) | 122 | 11
  Cycle 7, Week 1, Day 1 change from BL | -0.22 (1.882) | 0.06 (2.570)
  Cycle 8, Week 1, Day 1 change from BL: number analyzed (Participants) | 86 | 5
  Cycle 8, Week 1, Day 1 change from BL | 0.18 (1.926) | -0.26 (1.291)
  Cycle 9, Week 1, Day 1 change from BL: number analyzed (Participants) | 55 | 6
  Cycle 9, Week 1, Day 1 change from BL | -0.15 (1.751) | 0.12 (1.667)
  Cycle 10, Week 1, Day 1 change from BL: number analyzed (Participants) | 33 | 2
  Cycle 10, Week 1, Day 1 change from BL | 0.62 (2.141) | 1.50 (1.313)
  Cycle 11, Week 1, Day 1 change from BL: number analyzed (Participants) | 12 | 2
  Cycle 11, Week 1, Day 1 change from BL | -0.06 (1.334) | 0.36 (4.748)
  Cycle 12, Week 1, Day 1 change from BL: number analyzed (Participants) | 4 | 0
  Cycle 12, Week 1, Day 1 change from BL | -0.89 (0.914) |
  Cycle 13, Week 1, Day 1 change from BL: number analyzed (Participants) | 1 | 0
  Cycle 13, Week 1, Day 1 change from BL | -0.43 (NA) — NA: Only one participant analyzed |
  End of Treatment (EoT) change from BL: number analyzed (Participants) | 165 | 88
  End of Treatment (EoT) change from BL | 0.73 (2.756) | 0.29 (2.385)

22. Secondary Outcome: Time to Worsening in FACT-P Total Score
Description: Time to worsening was defined as the time from randomization to the first occurring of a >=10 point decrease in FACT-P total score compared to baseline, clinical disease progression, or death.
Time Frame: as for outcome 15
Population: PFS-Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Months | 5.7 [4.8 to 6.6] | 2.2 [1.8 to 2.8]

23. Secondary Outcome: Change From Baseline in FACT-P (Functional Assessment of Cancer Therapy - Prostate) Total Score
Description: The FACT-P total score (range 0-156) consist of five subscales (Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24)) and a functional well-being and prostate cancer subscale (range 0-48). Higher scores indicate higher degree of functioning and better quality of life.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Score on a scale
  Cycle 2, Week 1, Day 1 change from BL: number analyzed (Participants) | 304 | 100
  Cycle 2, Week 1, Day 1 change from BL | 3.6 (16.63) | -7.2 (17.85)
  Cycle 3, Week 1, Day 1 change from BL: number analyzed (Participants) | 269 | 52
  Cycle 3, Week 1, Day 1 change from BL | 3.8 (17.48) | -2.6 (14.00)
  Cycle 4, Week 1, Day 1 change from BL: number analyzed (Participants) | 222 | 32
  Cycle 4, Week 1, Day 1 change from BL | 5.4 (15.93) | -1.3 (18.40)
  Cycle 5, Week 1, Day 1 change from BL: number analyzed (Participants) | 181 | 21
  Cycle 5, Week 1, Day 1 change from BL | 4.0 (16.24) | -5.9 (27.83)
  Cycle 6, Week 1, Day 1 change from BL: number analyzed (Participants) | 158 | 13
  Cycle 6, Week 1, Day 1 change from BL | 4.1 (15.22) | -5.0 (26.87)
  Cycle 7, Week 1, Day 1 change from BL: number analyzed (Participants) | 122 | 11
  Cycle 7, Week 1, Day 1 change from BL | 4.9 (16.47) | -2.9 (17.89)
  Cycle 8, Week 1, Day 1 change from BL: number analyzed (Participants) | 86 | 5
  Cycle 8, Week 1, Day 1 change from BL | 3.8 (15.87) | -13.0 (32.76)
  Cycle 9, Week 1, Day 1 change from BL: number analyzed (Participants) | 54 | 6
  Cycle 9, Week 1, Day 1 change from BL | 3.8 (14.22) | 6.9 (5.92)
  Cycle 10, Week 1, Day 1 change from BL: number analyzed (Participants) | 33 | 2
  Cycle 10, Week 1, Day 1 change from BL | 0.0 (18.27) | 0.2 (14.14)
  Cycle 11, Week 1, Day 1 change from BL: number analyzed (Participants) | 12 | 2
  Cycle 11, Week 1, Day 1 change from BL | -0.8 (20.99) | 8.2 (33.71)
  Cycle 12, Week 1, Day 1 change from BL: number analyzed (Participants) | 4 | 0
  Cycle 12, Week 1, Day 1 change from BL | 10.3 (12.11) |
  Cycle 13, Week 1, Day 1 change from BL: number analyzed (Participants) | 1 | 0
  Cycle 13, Week 1, Day 1 change from BL | 30.0 (NA) — NA: Only one participant analyzed |
  End of Treatment (EoT) change from BL: number analyzed (Participants) | 161 | 86
  End of Treatment (EoT) change from BL | -9.4 (21.64) | -10.4 (18.59)

24. Secondary Outcome: Time to Worsening in EQ-5D-5L Utility Score
Description: Time to worsening for utility score was defined as time from randomization to the first occurrence of worsening in utility score relative to baseline (no change or any decrease), clinical disease progression, or death.
Time Frame: as for outcome 15
Population: PFS-Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Months | 1.0 [0.7 to 1.8] | 0.5 [0.4 to 1.0]

25. Secondary Outcome: Change From Baseline in the European Quality of Life (EuroQol) - 5 Domain 5 Level Scale (EQ-5D-5L) Utility Score
Description: The EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions. A utility score was obtained by using a weighted combination of the levels of the five dimension-scales. The weights were based on value sets which were country-specific for the U.K. Utility scores ranges from the lowest possible score for a living patient of -0.594 (when all responses are '5') to 1 (when all responses are '1').If a patient died, he was assigned a score of 0 on the date of death.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Score on a scale
  Cycle 2, Week 1, Day 1 change from BL: number analyzed (Participants) | 304 | 100
  Cycle 2, Week 1, Day 1 change from BL | 0.0221 (0.17693) | -0.0897 (0.24973)
  Cycle 3, Week 1, Day 1 change from BL: number analyzed (Participants) | 273 | 53
  Cycle 3, Week 1, Day 1 change from BL | 0.0297 (0.18817) | -0.0331 (0.14155)
  Cycle 4, Week 1, Day 1 change from BL: number analyzed (Participants) | 221 | 32
  Cycle 4, Week 1, Day 1 change from BL | 0.0292 (0.17713) | -0.0818 (0.23752)
  Cycle 5, Week 1, Day 1 change from BL: number analyzed (Participants) | 180 | 21
  Cycle 5, Week 1, Day 1 change from BL | 0.0398 (0.16827) | -0.0673 (0.28633)
  Cycle 6, Week 1, Day 1 change from BL: number analyzed (Participants) | 159 | 13
  Cycle 6, Week 1, Day 1 change from BL | 0.0342 (0.17950) | -0.0110 (0.17842)
  Cycle 7, Week 1, Day 1 change from BL: number analyzed (Participants) | 121 | 11
  Cycle 7, Week 1, Day 1 change from BL | 0.0252 (0.16127) | -0.0088 (0.09081)
  Cycle 8, Week 1, Day 1 change from BL: number analyzed (Participants) | 84 | 5
  Cycle 8, Week 1, Day 1 change from BL | 0.0285 (0.18017) | -0.0296 (0.14964)
  Cycle 9, Week 1, Day 1 change from BL: number analyzed (Participants) | 54 | 6
  Cycle 9, Week 1, Day 1 change from BL | 0.0100 (0.17447) | 0.0087 (0.08167)
  Cycle 10, Week 1, Day 1 change from BL: number analyzed (Participants) | 33 | 2
  Cycle 10, Week 1, Day 1 change from BL | 0.0134 (0.15764) | -0.0655 (0.09263)
  Cycle 11, Week 1, Day 1 change from BL: number analyzed (Participants) | 12 | 2
  Cycle 11, Week 1, Day 1 change from BL | 0.0464 (0.16858) | 0.0250 (0.19940)
  Cycle 12, Week 1, Day 1 change from BL: number analyzed (Participants) | 4 | 0
  Cycle 12, Week 1, Day 1 change from BL | 0.1118 (0.13833) |
  Cycle 13, Week 1, Day 1 change from BL: number analyzed (Participants) | 1 | 0
  Cycle 13, Week 1, Day 1 change from BL | 0.0640 (NA) — NA: Only one participant analyzed |
  End of Treatment (EoT) change from BL: number analyzed (Participants) | 163 | 85
  End of Treatment (EoT) change from BL | -0.0939 (0.22698) | -0.0900 (0.21223)

26. Secondary Outcome: Change From Baseline in the European Quality of Life (EuroQol) - 5 Domain 5 Level Scale (EQ-5D-5L) EQ-VAS
Description: The EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ VAS records the patient's self-rated health on a vertical visual analogue 0-100 scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The higher the EQ-VAS score, the better the QoL.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Score on a scale
  Cycle 2, Week 1, Day 1 change from BL: number analyzed (Participants) | 305 | 100
  Cycle 2, Week 1, Day 1 change from BL | 1.8 (19.98) | -7.2 (20.31)
  Cycle 3, Week 1, Day 1 change from BL: number analyzed (Participants) | 272 | 53
  Cycle 3, Week 1, Day 1 change from BL | 1.4 (19.82) | -3.8 (21.50)
  Cycle 4, Week 1, Day 1 change from BL: number analyzed (Participants) | 221 | 32
  Cycle 4, Week 1, Day 1 change from BL | 2.8 (19.18) | -1.7 (18.73)
  Cycle 5, Week 1, Day 1 change from BL: number analyzed (Participants) | 180 | 21
  Cycle 5, Week 1, Day 1 change from BL | 4.0 (17.30) | -8.5 (28.88)
  Cycle 6, Week 1, Day 1 change from BL: number analyzed (Participants) | 159 | 13
  Cycle 6, Week 1, Day 1 change from BL | 2.1 (19.61) | 3.2 (19.43)
  Cycle 7, Week 1, Day 1 change from BL: number analyzed (Participants) | 121 | 11
  Cycle 7, Week 1, Day 1 change from BL | 3.6 (20.64) | 5.9 (12.79)
  Cycle 8, Week 1, Day 1 change from BL: number analyzed (Participants) | 84 | 5
  Cycle 8, Week 1, Day 1 change from BL | 0.6 (17.18) | 13.8 (16.60)
  Cycle 9, Week 1, Day 1 change from BL: number analyzed (Participants) | 54 | 6
  Cycle 9, Week 1, Day 1 change from BL | 0.1 (19.68) | 6.3 (20.82)
  Cycle 10, Week 1, Day 1 change from BL: number analyzed (Participants) | 33 | 2
  Cycle 10, Week 1, Day 1 change from BL | 2.9 (13.97) | -8.0 (2.83)
  Cycle 11, Week 1, Day 1 change from BL: number analyzed (Participants) | 12 | 2
  Cycle 11, Week 1, Day 1 change from BL | 5.8 (10.33) | -9.0 (28.28)
  Cycle 12, Week 1, Day 1 change from BL: number analyzed (Participants) | 4 | 0
  Cycle 12, Week 1, Day 1 change from BL | 4.5 (13.03) |
  Cycle 13, Week 1, Day 1 change from BL: number analyzed (Participants) | 1 | 0
  Cycle 13, Week 1, Day 1 change from BL | -5.0 (NA) — NA: Only one participant analyzed |
  End of Treatment (EoT) change from BL: number analyzed (Participants) | 163 | 86
  End of Treatment (EoT) change from BL | -8.9 (22.07) | -10.1 (21.49)

27. Secondary Outcome: Number of Participants Hospitalized as In-patient
Description: The number of hospitalizations (yes/no) (admitted as in-patient) was collected as part of the hospital admission for health economic evaluations.
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Participants
  Yes | 157 | 59
  No | 228 | 137

28. Secondary Outcome: Duration of Time in Hospital Following 177Lu-PSMA-617 Administration
Description: The duration of time in hospital following 177Lu-PSMA-617 administration (hours) was the time span of patient discharged as captured on the 177Lu-PSMA-617 administration Case Report Form (CRF).
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 341 | 0
Hours | 28.25 (46.578) |

29. Secondary Outcome: Concomitant Drug Use for Health Economics Analysis
Description: The list of concomitant drugs as captured on the concomitant medication/therapy CRF page to include in each category was pre-specified and flagged prior to the pre planned analyses. (1) Bisphosphonates (including but not limited to zoledronic acid, alendronic acid, etc.), denosumab, and other bone targeted therapies), (2) Corticosteroids for systemic use (3), Antifungals for systemic use (i.e. ketoconazole), (4) ESA (erythropoietin stimulating agents, i.e. epoetin alfa), (5) Granulocyte macrophage colony-stimulating factor (GM-CSF), (6) Novel androgen axis drugs (NAADs; i.e. enzalutamide, abiraterone, apalutamide), (7) Antiemetics and (8) Opioid analgesics use for cancer-related pain.
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Participants
  Bisphosphonates: Yes | 169 | 88
  Bisphosphonates: No | 216 | 108
  Corticosteroids: Yes | 246 | 113
  Corticosteroids: No | 139 | 83
  Antifungals: Yes | 1 | 4
  Antifungals: No | 384 | 192
  Erythropoietin Stimulating Agents: Yes | 8 | 2
  Erythropoietin Stimulating Agents: No | 377 | 194
  Granulocyte macrophage colony-stimulating factor: Yes | 7 | 3
  Granulocyte macrophage colony-stimulating factor: No | 378 | 193
  Novel Androgen Axis Drugs: Yes | 188 | 115
  Novel Androgen Axis Drugs: No | 197 | 81
  Antiemetics: Yes | 232 | 45
  Antiemetics: No | 153 | 151
  Opioid analgesics: Yes | 199 | 96
  Opioid analgesics: No | 186 | 100

30. Secondary Outcome: Therapeutic Interventions for Health Economics Analysis
Description: The list of therapeutic interventions was pre-specified and flagged prior to the pre planned analyses as captured on: 1) the concurrent radiotherapy CRF page to include local external beam radiotherapy (inclusive of palliative external radiation), 2) on the concomitant medication/therapy CRF page to include blood transfusion (full blood or derivates).
Time Frame: as for outcome 9
Population: PFS Full Analysis Set (PFS-FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone
Number analyzed (Participants) | 385 | 196
Participants
  Local external beam therapy: Yes | 63 | 37
  Local external beam therapy: No | 322 | 159
  Blood transfusion: Yes | 74 | 13
  Blood transfusion: No | 311 | 183

31. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 30 days after last dose of study medication (on-treatment), up to approximately 43 months.
  Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approximately 66 months. These are not considered AEs
Time Frame: Pre-treatment deaths: Up to 28 days prior to treatment. On-treatment deaths: Up to approximately 43 months. Post-treatment deaths: Up to approximately 66 months
Population: Full Analysis Set (FAS) and the participants included in the sub-study.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC)
Number analyzed (Participants) | 551 | 280 | 30
Participants
  Pre-treatment deaths | 0 | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 529 | 205 | 30
  On-treatment deaths | 68 | 19 | 5
  Post-treatment deaths: number analyzed (Participants) | 461 | 186 | 25
  Post-treatment deaths | 389 | 182 | 16
  All deaths | 457 | 201 | 21

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 30 days post-treat follow-up, assessed up to approximately 43 months. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 66 months.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC): Main Study: 177Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC) - Events up to 30 days post-treatment
- Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone: Main Study: Best supportive/best standard of care (BS/BSOC) alone - Events up to 30 days post-treatment
- Main Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care(BS/BSOC): Main Study (Post-Treatment Survival Follow-Up): 177Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Main Study (Post-Tx Survival FU): Best Supportive/Best Standard of Care (BS/BSOC) Alone: Main Study (Post-Treatment Survival Follow-Up): Best supportive/best standard of care (BS/BSOC) alone - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Sub Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC): Sub Study (Post-Treatment Survival Follow-Up): 177Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC) - Deaths in the post-treatment survival follow-up were not considered adverse events.
Arm/Group | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) | Main Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care(BS/BSOC) | Main Study (Post-Tx Survival FU): Best Supportive/Best Standard of Care (BS/BSOC) Alone | Sub Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC)
All-Cause Mortality (participants affected / at risk) | 68/551 | 19/280 | 5/30 | 389/461 | 182/186 | 16/25
Serious Adverse Events (participants affected / at risk) | 195/529 | 58/205 | 9/30 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 502/529 | 151/205 | 28/30 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=529) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone (N=205) | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=30) | Main Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care(BS/BSOC) (N=0) | Main Study (Post-Tx Survival FU): Best Supportive/Best Standard of Care (BS/BSOC) Alone (N=0) | Sub Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=0)
Anaemia (Blood and lymphatic system disorders) | 15 | 1 | 2 | NA | NA | NA
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 6 | 0 | 0 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | NA | NA | NA
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | NA | NA | NA
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | NA | NA | NA
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 0 | NA | NA | NA
Vascular malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | NA | NA | NA
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | NA | NA | NA
Vision blurred (Eye disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 5 | 1 | 0 | NA | NA | NA
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0 | NA | NA | NA
Asthenia (General disorders) | 0 | 1 | 0 | NA | NA | NA
Disease progression (General disorders) | 2 | 1 | 0 | NA | NA | NA
Fatigue (General disorders) | 2 | 0 | 0 | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 1 | 1 | NA | NA | NA
Generalised oedema (General disorders) | 1 | 0 | 0 | NA | NA | NA
Influenza like illness (General disorders) | 0 | 1 | 0 | NA | NA | NA
Malaise (General disorders) | 1 | 0 | 0 | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | NA | NA | NA
Oedema (General disorders) | 0 | 1 | 0 | NA | NA | NA
Oedema peripheral (General disorders) | 1 | 0 | 0 | NA | NA | NA
Pain (General disorders) | 5 | 1 | 0 | NA | NA | NA
Pyrexia (General disorders) | 8 | 0 | 1 | NA | NA | NA
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | NA | NA | NA
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 2 | 0 | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Appendicitis (Infections and infestations) | 2 | 0 | 0 | NA | NA | NA
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Bronchitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
COVID-19 (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Extradural abscess (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Fungaemia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Infection (Infections and infestations) | 3 | 2 | 0 | NA | NA | NA
Kidney infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 7 | 3 | 0 | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 10 | 2 | 0 | NA | NA | NA
Septic shock (Infections and infestations) | 2 | 0 | 0 | NA | NA | NA
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 13 | 1 | 0 | NA | NA | NA
Urosepsis (Infections and infestations) | 3 | 0 | 0 | NA | NA | NA
Viral infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | NA | NA | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 2 | 0 | NA | NA | NA
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 5 | 1 | 1 | NA | NA | NA
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA | NA
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | NA | NA
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 3 | 1 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1 | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA | NA
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | NA | NA | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Cauda equina syndrome (Nervous system disorders) | 1 | 1 | 0 | NA | NA | NA
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Diplegia (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Hypoglossal nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 3 | 0 | 0 | NA | NA | NA
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Metabolic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | NA | NA | NA
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Pachymeningitis (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Paraplegia (Nervous system disorders) | 0 | 0 | 1 | NA | NA | NA
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Radiculopathy (Nervous system disorders) | 2 | 0 | 0 | NA | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Spinal cord compression (Nervous system disorders) | 6 | 11 | 0 | NA | NA | NA
Spinal cord disorder (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 4 | 0 | 0 | NA | NA | NA
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Tremor (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Confusional state (Psychiatric disorders) | 2 | 1 | 0 | NA | NA | NA
Delirium (Psychiatric disorders) | 1 | 1 | 0 | NA | NA | NA
Mental status changes (Psychiatric disorders) | 3 | 0 | 0 | NA | NA | NA
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0 | 0 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 10 | 6 | 0 | NA | NA | NA
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | NA | NA | NA
Haematuria (Renal and urinary disorders) | 11 | 1 | 0 | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | NA | NA | NA
Malignant urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 5 | 2 | 1 | NA | NA | NA
Urinary tract obstruction (Renal and urinary disorders) | 4 | 0 | 0 | NA | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | NA | NA | NA
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | NA | NA | NA
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Euthanasia (Surgical and medical procedures) | 1 | 0 | 0 | NA | NA | NA
Neck dissection (Surgical and medical procedures) | 1 | 0 | 0 | NA | NA | NA
Pain management (Surgical and medical procedures) | 1 | 0 | 0 | NA | NA | NA
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | NA | NA | NA
Embolism (Vascular disorders) | 2 | 0 | 0 | NA | NA | NA
Hypotension (Vascular disorders) | 4 | 0 | 0 | NA | NA | NA
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=529) | Main Study: Best Supportive/Best Standard of Care (BS/BSOC) Alone (N=205) | Sub Study: 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=30) | Main Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care(BS/BSOC) (N=0) | Main Study (Post-Tx Survival FU): Best Supportive/Best Standard of Care (BS/BSOC) Alone (N=0) | Sub Study (Post-Tx Survival FU): 177Lu-PSMA-617 Plus Best Supportive/Best Standard of Care (BS/BSOC) (N=0)
Anaemia (Blood and lymphatic system disorders) | 161 | 26 | 9 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 66 | 4 | 3 | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 75 | 8 | 5 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 45 | 3 | 0 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 91 | 9 | 4 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 30 | 6 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 103 | 23 | 3 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 101 | 5 | 3 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 205 | 1 | 5 | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 187 | 33 | 11 | NA | NA | NA
Toothache (Gastrointestinal disorders) | 4 | 0 | 2 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 97 | 12 | 4 | NA | NA | NA
Asthenia (General disorders) | 34 | 16 | 1 | NA | NA | NA
Extravasation (General disorders) | 0 | 0 | 2 | NA | NA | NA
Fatigue (General disorders) | 228 | 47 | 5 | NA | NA | NA
General physical health deterioration (General disorders) | 2 | 2 | 2 | NA | NA | NA
Oedema peripheral (General disorders) | 51 | 13 | 3 | NA | NA | NA
Pain (General disorders) | 28 | 10 | 2 | NA | NA | NA
Pyrexia (General disorders) | 30 | 7 | 1 | NA | NA | NA
Cystitis (Infections and infestations) | 6 | 0 | 2 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 54 | 1 | 1 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 38 | 12 | 0 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 20 | 2 | 2 | NA | NA | NA
Blood creatinine increased (Investigations) | 30 | 4 | 3 | NA | NA | NA
Weight decreased (Investigations) | 58 | 20 | 1 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 112 | 30 | 2 | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 36 | 7 | 1 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 39 | 7 | 0 | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 28 | 7 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 117 | 26 | 3 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 122 | 29 | 4 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 54 | 15 | 3 | NA | NA | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 12 | 2 | NA | NA | NA
Dizziness (Nervous system disorders) | 42 | 9 | 1 | NA | NA | NA
Headache (Nervous system disorders) | 36 | 4 | 2 | NA | NA | NA
Insomnia (Psychiatric disorders) | 28 | 9 | 2 | NA | NA | NA
Haematuria (Renal and urinary disorders) | 37 | 8 | 2 | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 8 | 4 | 3 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 13 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 19 | 2 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 2 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | NA | NA | NA
Hypertension (Vascular disorders) | 30 | 12 | 0 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03511664/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03511664/SAP_001.pdf